CLINICAL TRIAL: NCT05177107
Title: Phase 2b Randomized, Parallel, Double-blind, Placebo-Controlled, Repeat Dose, Multi-Site Study for Safety, Tolerability, and Efficacy of Personalized Phage Treatment and SoC for Subjects With Diabetic Foot Osteomyelitis Due to S. Aureus
Brief Title: Bacteriophage Therapy in Patients With Diabetic Foot Osteomyelitis
Acronym: DANCE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study reached minimum enrollment threshold
Sponsor: Adaptive Phage Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: APT.DFI.001
Record Dates: First submitted 2021-03-09; First posted 2022-01-04 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-01

CONDITIONS: Osteomyelitis; Diabetic Foot Osteomyelitis
Keywords: Diabetes; Osteomyelitis; Foot Infection; Phage Treatment; Bacteriophage; Phage; Bone Infection
MeSH Terms: conditions — Osteomyelitis; Diabetes Mellitus | interventions — Phage Therapy

STUDY DESIGN:
Intervention Model Description: 2:1, phage: placebo
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind:
  Patient will be randomized to receive either active phage or placebo treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1: Phage Therapy (Experimental): Bacteriophage therapy will be personalized for each patient dependent on phage susceptibility testing
  Interventions: Biological: Bacteriophage Therapy
- Group 2: Placebo (Placebo Comparator): Placebo (normal saline) will be administered using the same schedule and techniques as for Group 1 (phage therapy).
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Bacteriophage Therapy — Bacteriophage therapy will be personalized for each patient dependent on phage susceptibility testing
  Arms: Group 1: Phage Therapy
Other: Placebo — Placebo (normal saline)
  Arms: Group 2: Placebo

SUMMARY:
This is a phase 2b randomized trial designed to evaluate bacteriophage therapy in subjects with diabetic foot osteomyelitis.

DETAILED DESCRIPTION:
This study will evaluate the safety and efficacy of bacteriophage therapy in subjects with diabetic foot osteomyelitis (DFO). Enrolled subjects will have osteomyelitis infections due to Staph aureus. This study will include eligible subjects who have undergone or are planning to undergo surgical debridement of DFO.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 to <85 years of age.
* Ongoing diagnosis of diabetes.
* Have undergone or are scheduled to undergo surgical debridement for DFO as part of SoC, with the associated bone culture positive for S. aureus
* Availability of at least 1 matching phage for S. aureus cultured from the bone culture
* Receiving SoC treatment for DFO, including antibiotics after debridement and before randomization
* Meet defined study ulcer requirements as defined in the protocol
* Adequate circulation to the affected extremity demonstrated within 3 months prior to randomization and no revascularization procedure anticipated
* History of compliance with prior appointments and treatments in the investigator's opinion and willingness to receive and comply with SOC antimicrobial and clinical treatments for the study ulcer, including offloading

Exclusion Criteria:

* Healing of the ulcer by more than 30% between screening and randomization.
* Treated with hyperbaric oxygen or cellular/tissue products with 30 days of screening
* Suspicion of neoplasm associated with the study ulcer or any non-study diabetic ulcer independent of biopsy result.
* Presence of any cellulitis not localized to the study ulcer.
* Indwelling hardware at the site of the DFO.
* Body weight <50 kg.
* Presence of above ankle ulcer, with >50% above medial malleolus
* Hemoglobin < 7g/dL
* Abnormal liver function tests
* History of underlying liver disease at screening or within last 3 months
* Positive test for HIV-1 and /or HIV-2
* Any other clinically significant or severe disease that in the judgment of the investigator makes the patient unfit for the study or likely to withdraw prematurely from the study, or that could jeopardize the safety of the patient or confound the results of the study.
* Known allergy to phage products.
* Pregnant and/or breastfeeding.
* Immunocompromised at screening in the judgment of the investigator.
* Taking any systemic or topical antibacterial antibiotic within 2 weeks prior to the start of study treatment, for a condition other than Diabetic Foot Infection and DFO.
* Taking any antiviral medication within 2 weeks prior to the start of study treatment and up through the last administration of study treatment.
* Taking and/or receiving any therapies for the study ulcer that are not considered to be SOC.
* More than 30 days has elapsed between screening and randomization (start of treatment)
* Participating in another clinical trial within 4 weeks prior to screening.
* Inability to obtain or provide informed consent or adhere to the protocol in the judgment of the investigator.
* Once approximately 30% of subjects are enrolled with DFO involving digits, additional subjects will be excluded.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-11-24 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Percent area reduction of study ulcer through Week 13 | Baseline through Week 13
  Percent area reduction of the study ulcer surface area from baseline through Week 13

SECONDARY OUTCOMES:
Complete healing of the study ulcer | Baseline through Week 13
  Time to complete healing of the ulcer at any time point during the study
Time to 85% reduction of C-reactive protein (CRP) | Baseline through Week 13
  Time to 85% reduction of CRP at any time point during the study
Microbiological eradication of the target pathogen | baseline through Week 13
  Percentage of patients with microbiological eradication of the target pathogen at each time point during the study.

OTHER OUTCOMES:
Treatment-emergent AEs due to phage therapy | baseline through Week 12
  Number and percent of treatment-emergent Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Nitsan Halevy, MD, Principal Investigator — Medical Director
Locations (15):
- United States (15):
  - Southern Arizona VA Health Care System, Tuscon, Arizona
  - NorthBay Healthcare, Fairfield, California
  - Harbor Hospital / UCLA, Torrance, California
  - Rocky Mountain VA, Aurora, Colorado
  - Holy Cross Health, Fort Lauderdale, Florida
  - Infectious Disease Consultants od the Treasure Coast, Sebastian, Florida
  - Podiatry 1st / Gateway Clinical Trials, O'Fallon, Illinois
  - Foot & Ankle Center of Illinois, Springfield, Illinois
  - Henry Ford Health, Detroit, Michigan
  - Holy Name Medical Center, Teaneck, New Jersey
  - CurAlta Foot and Ankle, Westwood, New Jersey
  - Futuro Clinical Trials, LLC, McAllen, Texas
  - Bio X Cell Research LLC, San Antonio, Texas
  - Foot and Ankle Specialists of the Mid-Atlantic, Salem, Virginia
  - Salem VA, Salem, Virginia

IPD SHARING:
Plan to Share IPD: No